CLINICAL TRIAL: NCT01523067
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Response of Vasomera (PB1046) Injection Following a Single Subcutaneous Dose in Adult Subjects With Stage 1 or Stage 2 Essential Hypertension
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Response of Vasomera (PB1046) Injection Following a Single Subcutaneous Dose in Subjects With Stage 1 or 2 Essential Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0001
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Essential Hypertension
Keywords: Vasomera; PB1046; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — VIP-ELP fusion molecule PB1046; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasomera (PB1046) (Active Comparator)
  Interventions: Drug: Vasomera (PB1046)
- 0.9% Sodium Chloride (Placebo Comparator)
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Vasomera (PB1046) — Single dose of Vasomera
  Arms: Vasomera (PB1046)
Drug: 0.9% Sodium Chloride — Placebo injection
  Arms: 0.9% Sodium Chloride

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single ascending doses of Vasomera (PB1046) administered subcutaneously in adult subjects with Stage 1 or Stage 2 essential hypertension.

The secondary objectives of the study are to characterize the pharmacokinetic profile of single ascending doses of Vasomera and the relationship between serum concentrations of Vasomera and change in systolic and diastolic blood pressure as measured by:

* Mean change from baseline in 24-hour systolic and diastolic blood pressure measured by ambulatory blood pressure monitoring (ABPM) as compared to placebo.
* Identification of the minimum and maximum decrease in systolic and diastolic blood pressure as measured by ABPM.
* Mean change from baseline in cuff systolic and diastolic blood pressure as compared to placebo.
* Effect of Vasomera on pulse pressure and heart rate.

An additional secondary objective of this study will be to characterize the immunogenicity profile of Vasomera following a single subcutaneous dose.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study related procedures.
* Males or females age 18 - 70 years of age inclusive.
* Male and female subjects of childbearing potential must be willing and able to practice effective contraception during the study, and be willing and able to continue contraception for 1 month after their last dose of study drug.
* Diagnosis of essential hypertension and: Has a systolic blood pressure between 140-169 mmHg (between 130-169 mmHg if subject has type 2 diabetes mellitus (T2DM)) or diastolic blood pressure 90-109 mmHg (between 85 - 109 if subject has T2DM) who is not currently on antihypertensive therapy.
* or- Has been taking up to two antihypertensive agents to control blood pressure and who in the opinion of the investigator could be safely withdrawn from antihypertensive therapy.
* BMI ≥ 20 but ≤ 40 kg/m2
* The difference (highest to lowest mean values) in mean seated systolic blood pressure (triplicate measurements at 1-2 minute interval) measured on three separate occasions between Day -4 and Day 0 (pre-dose) is within 14 mmHg and diastolic is within 8 mmHg.
* Judged by the Investigator to be in generally stable health (except for hypertension) defined as absence of clinically significant laboratory abnormalities, vital signs, ECG findings or clinically significant underlying disease that would put the subject at risk for participation in the study, or would interfere with interpretation of the study results (i.e., secondary hypertension).
* Receiving stable doses of protocol permitted concomitant medications for 1 month prior to study drug administration with no anticipated dose adjustments during the study period.

Exclusion Criteria:

* Screening (triplicate sitting reading 1-2 minutes apart) BP > 169 mmHg (systolic) or > 109 mmHg (diastolic).
* Systolic blood pressure < 130 mmHg or > 169 mmHg and diastolic blood pressure < 85 mmHg or > 109 mmHg at randomization (Day -1) or prior to the first dose of study drug (Day 0)
* Unstable/underlying cardiovascular disease defined as in protocol.
* Uncontrolled type 2 diabetes mellitus defined as hemoglobin A1c > 9.0%
* Clinically significant renal and/or hepatic dysfunction at Screening or at baseline (Day -4) as defined in protocol.
* Use of non-steroidal anti-inflammatory drugs (excluding prophylactic use of low dose aspirin such as 81 - 162 mg) within 2 weeks prior to administration of study drug or anticipated use during the study period.
* Pregnant or lactating females.
* Known latex allergy (Ambulatory Blood Pressure Monitor [ABPM] unit contains latex in bladder and tubing).
* Known history of or active drug or alcohol abuse within the 12 months prior to Screening and/or positive drug screen or detection of alcohol at Screening or at baseline (Day -4).
* Positive for Human Immunodeficiency Virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies.
* Participation in any other study and have received any other investigational drug or device within 30 days prior to the Screening visit or are taking part in a non-drug study which in the opinion of the Investigator would interfere with the outcome of the study.
* Major surgery, donated or lost > or = 1 unit of blood (approximately 500 mL) within 1 month prior to randomization (Day -1) or display evidence of volume depletion (i.e., postural hypotension) not otherwise explained by the subject's antihypertensive medication regimen.
* Other medical or psychiatric condition which in the opinion of the Investigator would place the subject at increased risk, would preclude obtaining voluntary consent, or would interfere with the interpretation of the results of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability | Day -45 to Day 28
  * Incidence and severity of adverse events (AEs) and their relationship to Vasomera (including AEs of interest, gastrointestinal effects, injection site reaction and hypotension)
  * Changes in vital signs, ECGs, and safety laboratory parameters from baseline
  * Discontinuations from the study due to AEs

SECONDARY OUTCOMES:
Pharmacokinetics | Pre-dose, 1, 2, 3, 6, 8 and 12 hours post-dose, 24, 30 and 36 hours, Days 2, 3, 6, 7, 14, 21 and 28
  Maximum peak steady state drug concentration (Cmax), Time to Cmax (Tmax), Elimination Rate Constant, t1/2, AUC(inf), Total serum clearance, and Volume of distribution of Vasomera
Pharmacodynamics | ABPM (Day 0 and Day 6), Telemetry (Day -1, 0, 1 and Day 2 and 3 as needed), Daily home BP monitoring and Vital Signs (up to 3x times/day) during each visit (Day -35, -14, -7, -4, -1, 0, 1, 2, 3, 6, 7, 14, 21 and 28)
  * Change in mean 24-hour systolic blood pressure (SBP) and diastolic blood pressure (DBP) and mean daytime and mean nighttime SBP and DBP compared to placebo
  * Change in mean cuff systolic, diastolic and mean arterial blood pressure as compared to placebo
  * Mean change from baseline in effect of Vasomera on pulse pressure and heart rate
  * Proportion of subjects treated with study drug who were discontinued from treatment due to uncontrolled hypertension (i.e., SBP >169 mmHg or DBP >109 mmHg).
Immunogenicity | Pre-dose, Day 14 and Day 28
  Presence of anti-drug antibodies and anti-VIP antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Research
Locations (5):
- United States (5):
  - Pinnacle Research, Anniston, Alabama
  - Diablo Clinical Research, Walnut Creek, California
  - Prism Research Inc., Saint Paul, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Rainier Clinical Research, Renton, Washington